CLINICAL TRIAL: NCT05232773
Title: Rotator Cuff Surgery in Athletes: From Rehabilitation to Return to Sport
Acronym: RCR-SPORT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Silvia Sterzi, Full Professor, Campus Bio-Medico University
Other Study IDs: 62/21
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Rotator Cuff Tears; Athletes; Return to Sport
Keywords: Shoulder; Return to Sport; Rehabilitation; Athletes; Rotator Cuff; Rotator Cuff Injuries; Rotator Cuff Tears; Pilot Study; Assessment
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Enrolled patients will undergo supervised rehabilitation treatment for rotator cuff repair according to a standardized protocol (5 days/week) and will undergo clinical, kinematic and shoulder muscle strength assessments to collect data useful to define objective criteria for progression between rehabilitation phases. Assessment will be performed at four different times.
  The clinical evaluation of the shoulder is carried out through the Constant-Murley Score (CMS).
  Pain will be assessed through the visual analogical scale (VAS). Kinematic assessment (shoulder ROM, scapula-humeral rhythm, movement smoothness, movement speed) will be assessed through magneto-inertial measurements units (M-IMU).
  The maximal voluntary isometric contraction (MVIC) of shoulder flexor, abductor and rotator cuff muscles of the affected limb will be measured by the Chronojump Boscosystem® Force Sensor Kit
  Interventions: Procedure: Assessment
- Healthy subjects: Healthy subjects will undergo evaluations with the same timing as patients in the Experimental group.
  Interventions: Procedure: Assessment

INTERVENTIONS:
Procedure: Assessment — Evaluation of clinical and kinematic parameters

SUMMARY:
The main goal of this project is to study and define a rehabilitative flow-chart for athletes' rehabilitation and return to sport made by a set of objective shoulder evaluation indicators that are easy to use in clinical context. Enrolled patients will undergo supervised rehabilitation treatment for rotator cuff repair according to a standardized protocol (5 days/week) and will undergo four evaluation at different times. Healthy subjects will undergo evaluations with the same timing as patients.

DETAILED DESCRIPTION:
Clinical, kinematic and shoulder muscle strength assessments to collect data useful to define objective criteria for progression between rehabilitation phases will be performed according to the following times:

* T1 - 4-6 weeks after surgery: PROM assessment, pain assessment at rest and during PROM, Constant-Murley score (CMS).
* T2 - 6-12 weeks after surgery: AROM assessment (flexion in scapular plane, abduction, external and internal rotation), pain assessment at rest and during PROM and AROM tasks, scapular humeral rhythm, CMS.
* T3 - 12-16 weeks after surgery: AROM assessment (flexion in scapular plane, abduction, external and internal rotation), pain assessment at rest and during PROM and AROM tasks, scapular humeral rhythm, isometric strength assessment, CMS; joint proprioception assessment (joint position sense).
* T4 - 16-24 weeks after surgery: AROM assessment (flexion in scapular plane, abduction, external and internal rotation), scapular humeral rhythm, isometric strength assessment, CMS, joint proprioception assessment (joint position sense), movement speed and smoothness.

Enrolled patients will undergo supervised rehabilitation treatment for rotator cuff repair according to a standardized protocol (5 days/week) and will undergo the evaluations. Healthy subjects will undergo evaluations with the same timing as patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Mini Mental Status Examination (MMSE)> 24
* Acceptance and signature of informed consent

Exclusion Criteria:

* Presence of other pathologies that can compromise the standard post-operative course (shoulder instability; reoperation for failed rotator cuff repair; neurological and cognitive problems)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Competitive and non-competitive athletes undergoing rotator cuff repair surgery at the Unit of Orthopedics and Traumatology of the Campus Bio-Medico University Hospital will be considered eligible.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
To study and define a rehabilitative flow-chart for athletes' rehabilitation and return to sport | 2 years
  To create tool to support the multidisciplinary team involved in the decision-making process of progress between the various stages of rehabilitation and in the transition from the rehabilitation phase to the re-athletization phase after surgical repair of the rotator cuff of the shoulder in athletes

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Papalia, Professor, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Fondazione Policlinico Campus Bio-Medico, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided